CLINICAL TRIAL: NCT03249636
Title: Evaluation of New Markers for Minimal Residual Disease in Precursor B Acute Lymphoblastic Leukemia
Brief Title: New Markers for Minimal Residual Disease in Acute Lymphoblastic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maureen Farag, Principal Investigator, Assiut University
Other Study IDs: MFARAG
Record Dates: First submitted 2017-08-09; First posted 2017-08-15 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALL patients: New cases of patients with acute lymphocytic leukemia. Evaluation of markers 15 days after induction.
  Interventions: Diagnostic Test: Flow cytometric analysis

INTERVENTIONS:
Diagnostic Test: Flow cytometric analysis — Level of expression of the markers and the correlation between the markers with each other and with the clinical presentation and impact on patients with ALL.

SUMMARY:
Acute lymphoblastic leukemia , also known as acute lymphocytic leukemia, characterized by the overproduction and accumulation of cancerous, immature white blood cells, known as lymphoblasts, causing damage and death by inhibiting the production of normal cells (such as red and white blood cells and platelets) in the bone marrow and by spreading (infiltrating) to other organs. Acute lymphoblastic leukemia is most common in childhood, with a peak incidence at 2-5 years of age and another peak in old age.

DETAILED DESCRIPTION:
In recent years, new pieces of information obtained through immunophenotyping, cytogenetics and genomic profiling. Chemotherapy resistance have contributed to a better understanding of the pathology of this complex disorder and to recognition of subgroups of patients who respond differently to therapy.

The possible impact of the expression of various markers has been studied in ALL.

In patients with acute leukemia, treatment decisions are based on the status of peripheral blood and bone marrow cellularity. This provides a measure of the efficacy of therapy and can reveal leukemia relapse. The reliability of morphologic examination of peripheral blood and bone marrow largely depends on the hematologist's expertise, and its sensitivity is fundamentally limited by the similarities in appearance between leukemic cells and normal lympho-hematopoietic progenitors. Therefore, patients in complete morphologic remission may still have a large number of residual leukemic cells (potentially up to 1010).

Minimal residual disease (MRD) is currently the most powerful prognostic indicator in Precursor B acute lymphoblastic leukemia (B ALL). MRD analysis can be done by either ﬂow cytometric or molecular techniques. Flow cytometric detection holds potential for wider applicability than molecular techniques because ﬂow cytometric methods for leukemia diagnosis are already established at most cancer centers worldwide.

Flow cytometric detection of MRD is based on the principle that ALL cells express immunophenotypic features that can be used to distinguish them from normal hematopoietic cells, including hematogones and activated lymphocytes commonly referred to as Leukemia associated immunophenotype (LAIP). In virtually all patients with ALL, leukemia-associated immunophenotypes can be deﬁned at diagnosis and then used to monitor MRD during treatment.

The reliability of ﬂow cytometric MRD assays depends on several factors. The most important being the correct marker combination in use. Applicability is limited in some cases by the lack of suitable leukemia associated immunophenotype (LAIP) with the currently used markers and also antigen immunomodulation post treatment. Therefore, the identiﬁcation of new leukemia markers that are easily detectable and are stably expressed in a large proportion of ALL cases should simplify the application of MRD studies, help extend their beneﬁt to all patients and possibly enhance the sensitivity of MRD detection.

ELIGIBILITY:
Inclusion Criteria:

* 1. New cases of patients with acute lymphocytic leukemia. 2. Evaluation of markers 15 days after induction.

Exclusion Criteria:

* Patients died after induction
* Patients diagnosed as Non Hodgkin Lymphoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: New cases of patients with acute lymphocytic leukemia.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Level of expression of markers in acute lymphoblastic leukemia. | 1 year
  Level of expression of CD66c, CD 123 & CD 73 in acute lymphocytic leukemia ,the correlation with each other .and with the clinical assessment of patients before and after induction

CONTACTS AND LOCATIONS:
Overall Officials: Maureen R Farag, Resident, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Campana D, Coustan-Smith E. Measurements of treatment response in childhood acute leukemia. Korean J Hematol. 2012 Dec;47(4):245-54. doi: 10.5045/kjh.2012.47.4.245. Epub 2012 Dec 24. PMID 23320002
- [Background] Campana D, Behm FG. Immunophenotyping of leukemia. J Immunol Methods. 2000 Sep 21;243(1-2):59-75. doi: 10.1016/s0022-1759(00)00228-3. PMID 10986407
- [Background] Inaba H, Greaves M, Mullighan CG. Acute lymphoblastic leukaemia. Lancet. 2013 Jun 1;381(9881):1943-55. doi: 10.1016/S0140-6736(12)62187-4. Epub 2013 Mar 22. PMID 23523389